CLINICAL TRIAL: NCT04379726
Title: Characterization of β-cell Function and Insulin Sensitivity in Pre-transplant Patients With Cystic Fibrosis
Brief Title: β-cell Function and Insulin Sensitivity in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Emanuela Orsi, Head of Diabetology, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: FCMilano
Record Dates: First submitted 2020-04-28; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis-related Diabetes
Keywords: insulin; beta cell function; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with CFRD: Patients with diagnosis of CFRD, after OGTT
  Interventions: Behavioral: therapeutic optimization
- patients without CFRD: Patients without diagnosis of CFRD, after OGTT

INTERVENTIONS:
Behavioral: therapeutic optimization — patients with diagnosis of CFRD will undergo the gold standard treatment for the disease (insulin therapy)
  Groups: patients with CFRD

SUMMARY:
Cystic fibrosis is a genetic disorder caused by mutations in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gene, leading to pulmonary infections, sinus disease, pancreatic insufficiency, hepatobiliary disease and male infertility, with respiratory failure being the primary cause of death. Cystic Fibrosis Related Diabetes (CFRD) in one of the most common complication of cystic fibrosis (CF) and it's associated with a worse respiratory and nutritional state, with a negative impact on life expectancy. It differs from type 1 diabetes and type 2 diabetes for particular characteristics making this disease a separated clinical entity.

To date, there is a lack of evidence on many aspects concerning this disease:

* the pathophysiology of the disease: decreased insulin secretion has historically been seen has the major trigger for CFRD, but data about this mechanism are scarce and conflicting. Moreover, the role of insulin-resistance seems to be not consistent, but pulmonary exacerbations are very common and, in this setting, insulin sensitivity can worsen significantly.
* the relationship between its development and particular genetic settings: certain CFTR genotypes are known to be most related to the risk of diabetes, and only few susceptibility genes for type 2 diabetes have been evaluated as potential predisposing factors for CFRD.
* the relationship between the therapeutic optimization and its impact on metabolic status and lung function: CFRD is known to be associated with worse clinical outcomes, reflected in more frequent clinical exacerbations, greater reduction in lung function, poorer nutritional status and decreased survival. It has also been demonstrated that insulin therapy can improve pulmonary function, increase body weight and reduce lung exacerbations. However, no study on the clinical impact of the optimization of insulin therapy on pulmonary outcomes and life expectancy are available in this population.
* finally, no data about potential predisposing pre-transplant risk factors for development of post-transplant DM are available

For this reason, the investigators have structured a study with the aim to:

* characterize the pathophysiological process leading to CFRD, with assessment of the relative contribution of the insulin resistance and the β-cellular secretion impairment
* define the prevalence of CFRD in relation to the mutations of the CFTR gene and to the presence of candidate genes for the development of type 2 diabetes
* perform a proteomic analysis to identify potential proteomic biomarkers among CFRD patients
* evaluate the body composition, muscle performance and respiratory outcomes in patients on insulin therapy, before and after therapeutic optimization, in a follow-up period of 24 months.
* identify eventual predisposing factors for the development of post-transplant diabetes in subjects without pre-transplant CFRD.

DETAILED DESCRIPTION:
The study aims are:

* Task 1: pathophysiological characterization of CFRD with assessment of the relative contribution of the insulin resistance and the β-cellular secretion impairment through the use of a Minimum Model applied to OGTT for the evaluation of insulin sensitivity and secretion
* Task 2:

  2a) determination of the prevalence of CFRD in relation to the mutations of the CFTR gene (presence of mutations with residual function of the CFTR protein) 2b) determination of the prevalence of CFRD in relation to the presence of candidate genes for the devel-opment of type 2 diabetes (NOTCH2, BCL11A, THADA, IGFBP-2, PPARG, ADAMTS9, CDKAL1, VEFGA, JAZF1, CDKN2A / 2B, HHEX, CDC123 / CAMK1D, TCF7L2, KCNJ11, DCD, TSPAN8 / LGR5, FTO, WFS1, SLC30A8 and INS).

  2c) determination of variations in the proteomic analysis of CFRD patients compared to CF without DM and a control group of healthy individuals.
* Task 3: evaluation of the effect of the therapeutic optimization of glycometabolic control on body composition and respiratory outcomes in patients on insulin therapy, in a follow-up period of 24 months.
* Task 4: identification of predisposing factors for the development of post-transplant diabetes in subjects without CFRD.

METHODS:

All CF patients currently followed at the Unit of Pulmonology of our Center (250 subjects) will be considered eligible for the study.

Total duration of the study: 156 weeks (3 years).

The enrolled patients will be divided into two groups:

GROUP 1: subjects with a negative history for CFRD or with a CFRD diagnosis that does not require insulin therapy GROUP 2: subjects suffering from CFRD in insulin therapy

Protocol 1: Group 1; metabolic and anthropometric evaluation and assessment of insulin sensitivity / secretion.

Protocol 2: Group 1 and Group 2; genetic evaluation / proteomic evaluation Protocol 3: Group 2; pre- and post-intervention metabolic, anthropometric and nutritional assessment.

Protocol 4: Group 1 patients without CFRD undergoing lung transplantation (10); genetic, metabolic, an-thropometric and pre-and post-transplant assessment of insulin sensitivity / secretion.

Patients will undergo a:

1. METABOLIC EVALUATION: a venous sampling will be performed for blood glucose, HbA1c, total cholesterol, HDL, triglycerides, blood count, albumin, total proteins, pseudocholinesterase, AST, ALT, GGT, ALP, 25OHvitD
2. GENETIC EVALUATION: the investigators will evaluate the specific genetic mutation of the CFTR gene and the presence of gene variants related to the development of DM2 (NOTCH2, BCL11A, THADA, IGFBP-2, PPARG, ADAMTS9, CDKAL1, VEFGA, JAZF1, CDKN2A / 2B, HHEX, CDC123 / CAMK1D, TCF7L2, KCNJ11, DCD, TSPAN8 / LGR5, FTO, WFS1, SLC30A8 and INS)
3. PROTEOMIC EVALUATION: the investigators will perform a Mass Spectrometry to identify variations in the protein pattern expression in CFRD patients if compared to CF patients without DM and healthy control individuals. The list of analyzed protein is available in supplemental data 2.
4. ANTROPOMETRIC EVALUATION. the anthropometric evaluation will be performed with objective exami-nation (Body Mass Index - BMI, waist circumference - CV and hip circumference - CF) , DEXA total body and bioimpedentiometry
5. DYNAMIC EVALUATION OF INSULIN SENSITIVITY AND β CELL SECRETION. Patients will undergo a 5-hours OGTT with serial blood samples and with the application of a Mathematical Model adapted ad hoc (Appendix 1 for a detailed description of the model), in order to quantify the contribution of insulin resistance and β-cell secretion to the development of CFRD
6. PULMONARY EVALUATION. According to clinical practice, patients will be subjected to respiratory function tests with the calculation of FEV1 (absolute and percentage), exacerbation rate, rate of severe exacerbation (need of hospitalization), patient-reported outcomes (PROs) obtained from the sCF-quality of life questionnaire, which will be provided to patients in paper form.

SAMPLE SIZE AND STATISTICAL ANALYSIS:

Referring to the primary objective of the project, the observational nature of the study and the absence of evidence about the topic make a precise evaluation of the power of the study a difficult issue. However, considering the number of patients available and followed by our Center (n = 136), it has been calculated that the present study will have the power of 80% and an alpha level equal to 5% to show a significant reduction of at least 25% in the 1st phase secretion in the group of diabetics if compared to the non-diabetic group (assuming a mean value in non-diabetics of 1500 (aggiungere udm) and a SD of 500 (udm) (Pass v. 11 NCSS software, LCC, Kaysville, Utah, USA).

A series of descriptive analyzes will be performed: the continuous variables will be presented as averages and standard deviations or median with interquartile ranges, depending on the distribution. Frequency distributions will be presented as numbers and percentages. Data will also be presented graphically with histograms and "Box-and-Whisker" plots in order to evaluate potential anomalous values, allowing a further data-check phase in order to have reliable data for subsequent analyzes. Differences between the groups will be analyzed using parametric tests (t-test or ANOVA) without repeated tests or repeated tests, depending on the task of the project. If the normality of the distributions were violated (normal test based on the Shapiro-Wilk statistics), non-parametric technical correspondents will be used. Categorical data will be compared using contingency tables through the Chi-square test or Fisher's exact test, where appropriate. All tests will be two-tailed and p-values less than 5% will be considered statistically significant.

A series of descriptive analyzes will be performed: the continuous variables will be presented as averages and standard or median deviations with interquartile ranges, depending on the distribution. Frequency distributions will be presented as numbers and percentages. The data will also be presented graphically through histograms and "Box-and-Whisker" plots in order to evaluate potential anomalous values that will allow a further data-check phase in order to have valid data for subsequent analyzes. The differences between the groups will be analyzed using parametric techniques (t-test or ANOVA) without repeated tests or with repeated tests, depending on the task of the project. If the normality of the distributions was violated (normality test based on the Shapiro-Wilk statistics), corresponding non-parametric techniques will be used. Categorical data will be compared using contingency tables through the Chi-square test or Fisher's exact test, where appropriate. All tests will be two-tailed and a p-values less than 5% will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* written informed
* diagnosis of cystic fibrosis

Exclusion Criteria:

* celiac disease
* pregnancy
* diagnosis of T1DM

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients will be followed for three years as described in the protocol
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
TASK 1: derivative control (DC) | 2 YEARS
  index of first phase insulin secretion, calculated using the Minimum Model applied to the OGTT in patients with CF and various degrees of glucose homeostasis
TASK 1: proportional control (PC) | 2 YEARS
  index of second phase insulin secretion, calculated using the Minimum Model applied to the OGTT in patients with CF and various degrees of glucose homeostasis
TASK 1: OGIS-2H | 2 YEARS
  index of insulin sensitivity, calculated with the appropriate formula applied to the OGTT in patients with CF and various degrees of glucose homeostasis
TASK 2: prevalence of CFRD in relation to the classes of mutations in the CFTR gene | 2 YEARS
TASK 3: variation of FEV1 | 2 YEARS
  difference between pre- and post-institution of an optimal glycemic control
TASK 4: incidence of post-transplant diabetes in subjects without CFRD | 2 YEARS

SECONDARY OUTCOMES:
TASK 2: prevalence of candidate genes for DM2 in the population with CF | 2 YEARS
TASK2: variations in the protein pattern expression in CFRD population | 2 YEARS
  highlighted with a proteomic analysis
TASK 3: variations of other respiratory and muscle-performance parameters | 2 YEARS
  n° episodes of exacerbation/year, n° of severe exacerbation (need of hospitalization)/year, and patient-reported outcomes (PROs) obtained from a specific validated questionnaire (CF-quality of life questionnaire, 9 quality of life domains: Physical Functioning, Vitality, Emotional state, Social limitations, Role Limitations/School Performance, Embarrassment, Body Image, Eating Disturbances, Treatment Constraints. 3 symptom scales: Respiratory, Digestive, Weight. 1 health perception scale: Health Status (present/evolution).Scores range from 0 to 100, with higher scores indicating better health)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacKenzie T, Gifford AH, Sabadosa KA, Quinton HB, Knapp EA, Goss CH, Marshall BC. Longevity of patients with cystic fibrosis in 2000 to 2010 and beyond: survival analysis of the Cystic Fibrosis Foundation patient registry. Ann Intern Med. 2014 Aug 19;161(4):233-41. doi: 10.7326/M13-0636. PMID 25133359
- [Result] Yoon JC. Evolving Mechanistic Views and Emerging Therapeutic Strategies for Cystic Fibrosis-Related Diabetes. J Endocr Soc. 2017 Oct 30;1(11):1386-1400. doi: 10.1210/js.2017-00362. eCollection 2017 Nov 1. PMID 29264462
- [Result] Haardt M, Benharouga M, Lechardeur D, Kartner N, Lukacs GL. C-terminal truncations destabilize the cystic fibrosis transmembrane conductance regulator without impairing its biogenesis. A novel class of mutation. J Biol Chem. 1999 Jul 30;274(31):21873-7. doi: 10.1074/jbc.274.31.21873. PMID 10419506
- [Result] Rowe SM, Miller S, Sorscher EJ. Cystic fibrosis. N Engl J Med. 2005 May 12;352(19):1992-2001. doi: 10.1056/NEJMra043184. No abstract available. PMID 15888700
- [Result] Moran A, Dunitz J, Nathan B, Saeed A, Holme B, Thomas W. Cystic fibrosis-related diabetes: current trends in prevalence, incidence, and mortality. Diabetes Care. 2009 Sep;32(9):1626-31. doi: 10.2337/dc09-0586. Epub 2009 Jun 19. PMID 19542209
- [Result] Marshall BC, Butler SM, Stoddard M, Moran AM, Liou TG, Morgan WJ. Epidemiology of cystic fibrosis-related diabetes. J Pediatr. 2005 May;146(5):681-7. doi: 10.1016/j.jpeds.2004.12.039. PMID 15870674
- [Result] Blackman SM, Tangpricha V. Endocrine Disorders in Cystic Fibrosis. Pediatr Clin North Am. 2016 Aug;63(4):699-708. doi: 10.1016/j.pcl.2016.04.009. PMID 27469183
- [Result] Blackman SM, Commander CW, Watson C, Arcara KM, Strug LJ, Stonebraker JR, Wright FA, Rommens JM, Sun L, Pace RG, Norris SA, Durie PR, Drumm ML, Knowles MR, Cutting GR. Genetic modifiers of cystic fibrosis-related diabetes. Diabetes. 2013 Oct;62(10):3627-35. doi: 10.2337/db13-0510. Epub 2013 May 13. PMID 23670970
- [Result] Lewis C, Blackman SM, Nelson A, Oberdorfer E, Wells D, Dunitz J, Thomas W, Moran A. Diabetes-related mortality in adults with cystic fibrosis. Role of genotype and sex. Am J Respir Crit Care Med. 2015 Jan 15;191(2):194-200. doi: 10.1164/rccm.201403-0576OC. PMID 25479583
- [Result] Adler AI, Shine BS, Chamnan P, Haworth CS, Bilton D. Genetic determinants and epidemiology of cystic fibrosis-related diabetes: results from a British cohort of children and adults. Diabetes Care. 2008 Sep;31(9):1789-94. doi: 10.2337/dc08-0466. Epub 2008 Jun 5. PMID 18535191
- [Result] Milla CE, Warwick WJ, Moran A. Trends in pulmonary function in patients with cystic fibrosis correlate with the degree of glucose intolerance at baseline. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):891-5. doi: 10.1164/ajrccm.162.3.9904075. PMID 10988101
- [Result] Schaedel C, de Monestrol I, Hjelte L, Johannesson M, Kornfalt R, Lindblad A, Strandvik B, Wahlgren L, Holmberg L. Predictors of deterioration of lung function in cystic fibrosis. Pediatr Pulmonol. 2002 Jun;33(6):483-91. doi: 10.1002/ppul.10100. PMID 12001283
- [Result] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Result] Smyth AR, Bell SC, Bojcin S, Bryon M, Duff A, Flume P, Kashirskaya N, Munck A, Ratjen F, Schwarzenberg SJ, Sermet-Gaudelus I, Southern KW, Taccetti G, Ullrich G, Wolfe S; European Cystic Fibrosis Society. European Cystic Fibrosis Society Standards of Care: Best Practice guidelines. J Cyst Fibros. 2014 May;13 Suppl 1:S23-42. doi: 10.1016/j.jcf.2014.03.010. PMID 24856775
- [Result] Lanng S, Thorsteinsson B, Roder ME, Nerup J, Koch C. Insulin sensitivity and insulin clearance in cystic fibrosis patients with normal and diabetic glucose tolerance. Clin Endocrinol (Oxf). 1994 Aug;41(2):217-23. doi: 10.1111/j.1365-2265.1994.tb02533.x. PMID 7923827
- [Result] Kelly A, Moran A. Update on cystic fibrosis-related diabetes. J Cyst Fibros. 2013 Jul;12(4):318-31. doi: 10.1016/j.jcf.2013.02.008. Epub 2013 Apr 3. PMID 23562217
- [Result] Moran A, Diem P, Klein DJ, Levitt MD, Robertson RP. Pancreatic endocrine function in cystic fibrosis. J Pediatr. 1991 May;118(5):715-23. doi: 10.1016/s0022-3476(05)80032-0. PMID 2019925
- [Result] Sheikh S, Gudipaty L, De Leon DD, Hadjiliadis D, Kubrak C, Rosenfeld NK, Nyirjesy SC, Peleckis AJ, Malik S, Stefanovski D, Cuchel M, Rubenstein RC, Kelly A, Rickels MR. Reduced beta-Cell Secretory Capacity in Pancreatic-Insufficient, but Not Pancreatic-Sufficient, Cystic Fibrosis Despite Normal Glucose Tolerance. Diabetes. 2017 Jan;66(1):134-144. doi: 10.2337/db16-0394. Epub 2016 Aug 5. PMID 27495225
- [Result] Moran A, Doherty L, Wang X, Thomas W. Abnormal glucose metabolism in cystic fibrosis. J Pediatr. 1998 Jul;133(1):10-17. doi: 10.1016/s0022-3476(98)70171-4. No abstract available. PMID 9672504
- [Result] Ode KL, Moran A. New insights into cystic fibrosis-related diabetes in children. Lancet Diabetes Endocrinol. 2013 Sep;1(1):52-8. doi: 10.1016/S2213-8587(13)70015-9. Epub 2013 May 23. PMID 24622267
- [Result] Koivula FNM, McClenaghan NH, Harper AGS, Kelly C. Islet-intrinsic effects of CFTR mutation. Diabetologia. 2016 Jul;59(7):1350-1355. doi: 10.1007/s00125-016-3936-1. Epub 2016 Mar 31. PMID 27033560
- [Result] Guo JH, Chen H, Ruan YC, Zhang XL, Zhang XH, Fok KL, Tsang LL, Yu MK, Huang WQ, Sun X, Chung YW, Jiang X, Sohma Y, Chan HC. Glucose-induced electrical activities and insulin secretion in pancreatic islet beta-cells are modulated by CFTR. Nat Commun. 2014 Jul 15;5:4420. doi: 10.1038/ncomms5420. PMID 25025956
- [Result] Ali BR. Is cystic fibrosis-related diabetes an apoptotic consequence of ER stress in pancreatic cells? Med Hypotheses. 2009 Jan;72(1):55-7. doi: 10.1016/j.mehy.2008.07.058. Epub 2008 Oct 11. PMID 18851900
- [Result] Hudson VM. Rethinking cystic fibrosis pathology: the critical role of abnormal reduced glutathione (GSH) transport caused by CFTR mutation. Free Radic Biol Med. 2001 Jun 15;30(12):1440-61. doi: 10.1016/s0891-5849(01)00530-5. PMID 11390189
- [Result] Ntimbane T, Comte B, Mailhot G, Berthiaume Y, Poitout V, Prentki M, Rabasa-Lhoret R, Levy E. Cystic fibrosis-related diabetes: from CFTR dysfunction to oxidative stress. Clin Biochem Rev. 2009 Nov;30(4):153-77. PMID 20011209
- [Result] Edlund A, Esguerra JL, Wendt A, Flodstrom-Tullberg M, Eliasson L. CFTR and Anoctamin 1 (ANO1) contribute to cAMP amplified exocytosis and insulin secretion in human and murine pancreatic beta-cells. BMC Med. 2014 May 28;12:87. doi: 10.1186/1741-7015-12-87. PMID 24885604
- [Result] Edlund A, Pedersen MG, Lindqvist A, Wierup N, Flodstrom-Tullberg M, Eliasson L. CFTR is involved in the regulation of glucagon secretion in human and rodent alpha cells. Sci Rep. 2017 Mar 7;7(1):90. doi: 10.1038/s41598-017-00098-8. PMID 28273890
- [Result] Sun X, Yi Y, Xie W, Liang B, Winter MC, He N, Liu X, Luo M, Yang Y, Ode KL, Uc A, Norris AW, Engelhardt JF. CFTR Influences Beta Cell Function and Insulin Secretion Through Non-Cell Autonomous Exocrine-Derived Factors. Endocrinology. 2017 Oct 1;158(10):3325-3338. doi: 10.1210/en.2017-00187. PMID 28977592
- [Result] Farrell PM, White TB, Ren CL, Hempstead SE, Accurso F, Derichs N, Howenstine M, McColley SA, Rock M, Rosenfeld M, Sermet-Gaudelus I, Southern KW, Marshall BC, Sosnay PR. Diagnosis of Cystic Fibrosis: Consensus Guidelines from the Cystic Fibrosis Foundation. J Pediatr. 2017 Feb;181S:S4-S15.e1. doi: 10.1016/j.jpeds.2016.09.064. PMID 28129811
- [Result] Moran A, Pyzdrowski KL, Weinreb J, Kahn BB, Smith SA, Adams KS, Seaquist ER. Insulin sensitivity in cystic fibrosis. Diabetes. 1994 Aug;43(8):1020-6. doi: 10.2337/diab.43.8.1020. PMID 8039595
- [Result] Austin A, Kalhan SC, Orenstein D, Nixon P, Arslanian S. Roles of insulin resistance and beta-cell dysfunction in the pathogenesis of glucose intolerance in cystic fibrosis. J Clin Endocrinol Metab. 1994 Jul;79(1):80-5. doi: 10.1210/jcem.79.1.8027259.
- [Result] American Diabetes Association. 1. Improving Care and Promoting Health in Populations: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S7-S13. doi: 10.2337/dc20-S001. PMID 31862744
- [Result] Moran A, Pekow P, Grover P, Zorn M, Slovis B, Pilewski J, Tullis E, Liou TG, Allen H; Cystic Fibrosis Related Diabetes Therapy Study Group. Insulin therapy to improve BMI in cystic fibrosis-related diabetes without fasting hyperglycemia: results of the cystic fibrosis related diabetes therapy trial. Diabetes Care. 2009 Oct;32(10):1783-8. doi: 10.2337/dc09-0585. Epub 2009 Jul 10. PMID 19592632
- [Result] Dobson L, Hattersley AT, Tiley S, Elworthy S, Oades PJ, Sheldon CD. Clinical improvement in cystic fibrosis with early insulin treatment. Arch Dis Child. 2002 Nov;87(5):430-1. doi: 10.1136/adc.87.5.430. No abstract available. PMID 12390923
- [Result] Mozzillo E, Franzese A, Valerio G, Sepe A, De Simone I, Mazzarella G, Ferri P, Raia V. One-year glargine treatment can improve the course of lung disease in children and adolescents with cystic fibrosis and early glucose derangements. Pediatr Diabetes. 2009 May;10(3):162-7. doi: 10.1111/j.1399-5448.2008.00451.x. Epub 2009 Jan 14. PMID 19207231
- [Result] Grancini V, Trombetta M, Lunati ME, Zimbalatti D, Boselli ML, Gatti S, Donato MF, Resi V, D'Ambrosio R, Aghemo A, Pugliese G, Bonadonna RC, Orsi E. Contribution of beta-cell dysfunction and insulin resistance to cirrhosis-associated diabetes: Role of severity of liver disease. J Hepatol. 2015 Dec;63(6):1484-90. doi: 10.1016/j.jhep.2015.08.011. Epub 2015 Aug 20. PMID 26297917
- [Result] Bonadonna RC, Heise T, Arbet-Engels C, Kapitza C, Avogaro A, Grimsby J, Zhi J, Grippo JF, Balena R. Piragliatin (RO4389620), a novel glucokinase activator, lowers plasma glucose both in the postabsorptive state and after a glucose challenge in patients with type 2 diabetes mellitus: a mechanistic study. J Clin Endocrinol Metab. 2010 Nov;95(11):5028-36. doi: 10.1210/jc.2010-1041. Epub 2010 Aug 25. PMID 20739378
- [Result] Mari A, Pacini G, Murphy E, Ludvik B, Nolan JJ. A model-based method for assessing insulin sensitivity from the oral glucose tolerance test. Diabetes Care. 2001 Mar;24(3):539-48. doi: 10.2337/diacare.24.3.539. PMID 11289482
- [Result] Cobelli C, Toffolo GM, Dalla Man C, Campioni M, Denti P, Caumo A, Butler P, Rizza R. Assessment of beta-cell function in humans, simultaneously with insulin sensitivity and hepatic extraction, from intravenous and oral glucose tests. Am J Physiol Endocrinol Metab. 2007 Jul;293(1):E1-E15. doi: 10.1152/ajpendo.00421.2006. Epub 2007 Mar 6. PMID 17341552
- [Result] Mari A, Camastra S, Toschi E, Giancaterini A, Gastaldelli A, Mingrone G, Ferrannini E. A model for glucose control of insulin secretion during 24 h of free living. Diabetes. 2001 Feb;50 Suppl 1:S164-8. doi: 10.2337/diabetes.50.2007.s164. PMID 11272182
- [Derived] Grancini V, Alicandro G, Porcaro LL, Zazzeron L, Gramegna A, Morlacchi LC, Rossetti V, Gaglio A, Resi V, Dacco V, Blasi F, Orsi E. Effects of insulin therapy optimization with sensor augmented pumps on glycemic control and body composition in people with cystic fibrosis-related diabetes. Front Endocrinol (Lausanne). 2023 Aug 31;14:1228153. doi: 10.3389/fendo.2023.1228153. eCollection 2023. PMID 37720540
- See also: Related Info — http://cftr2.org